CLINICAL TRIAL: NCT01588418
Title: Effect of Exenatide on Brain Glucose Uptake in Relations to Pancreatic, Adipose Tissue, and Hepatic Function
Brief Title: Acute Effect of Exenatide on Brain Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Ralph DeFronzo, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 233-GAS-08
Record Dates: First submitted 2012-03-19; First posted 2012-05-01 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Impaired Glucose Tolerance (IGT); Diabetes
Keywords: Impaired glucose tolerance (IGT); Diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide first, then Placebo (Experimental): Exenatide 5mcg was injected subcutaneously 30 min before Oral Glucose Tolerance Test (OGTT)-PET study. The same subject was studied again a few weeks later with the same protocol with Placebo injection.
  Interventions: Drug: Exenatide; Drug: Placebo
- Placebo first, then Exenatide (Experimental): Placebo was injected subcutaneously 30 min before OGTT-PET study. The same subject was studied again a few weeks later with the same protocol with injection of Exenatide 5mcg .
  Interventions: Drug: Exenatide; Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide (5mcg) was administered in random order 30 min before OGTT-PET study, crossover study
  Other Names: Byetta
Drug: Placebo — Placebo was administered in random order 30 min before OGTT-PET study in the same subject

SUMMARY:
This research study will examine brain glucose metabolism after an overnight fast to determine the effect of exenatide on brain glucose metabolism and lipid metabolism.

DETAILED DESCRIPTION:
This study will elucidate if exenatide has an effect on brain glucose metabolism. This will be accomplished by measuring the rate of glucose binding in various brain regions by Positron Emission Tomography (PET) after glucose load with exenatide injection and compare it with placebo injection measured in the same subject. The changes will be compared with peripheral and hepatic glucose metabolism and lipolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males age 18-65 years old
2. Patients must have Body Mass Index (BMI) between 25 and 40 kg/m2
3. 2-hour glucose concentration above 140mg/dl after 75g glucose load, ie, having impaired glucose tolerance or newly diagnosed type 2 diabetes.
4. Patients must have BMI of 25-40 kg/m2
5. Patients must have no known severe liver or kidney disease, cancer, neurologic, psychiatric or systemic disease, ability to understand the study.
6. Only patients whose body weight has been stable (±3-4 pounds) over the three months prior to study will be included.
7. Patients must have the following laboratory values:

   * Hematocrit ≥ 34 vol%
   * Serum creatinine* ≤ 1.5 mg/dl in males and
   * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT): ≤ 2.5 times upper limit of normal
   * Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT): ≤ 2.5 times upper limit of normal
   * Alkaline phosphatase ≤ 2.5 times upper limit of normal
   * If serum creatinine is ≤ 1.5 mg/dl in males, the PI can grant an exception and not exclude the patient if the Glomerular filtration rate (GFR) is >70 ml/min

Exclusion Criteria:

Patients are excluded from participation in the study if they meet any of the following criteria:

1. Patients with major chronic illness (cancer, liver, kidney, cardiovascular disease)
2. Patients with BMI over 40 and under 25
3. Patient with age below 18 yrs and over 65 yrs
4. Female subjects
5. Patients with type 1 diabetes
6. Patients treated for type 2 diabetes
7. Subjects with normal glucose tolerance (NGT)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Gastaldelli, PhD, Principal Investigator — UTHSCSA, San Antonio, TX
Locations (1):
- Texas Diabetes Institute and UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daniele G, Iozzo P, Molina-Carrion M, Lancaster J, Ciociaro D, Cersosimo E, Tripathy D, Triplitt C, Fox P, Musi N, DeFronzo R, Gastaldelli A. Exenatide Regulates Cerebral Glucose Metabolism in Brain Areas Associated With Glucose Homeostasis and Reward System. Diabetes. 2015 Oct;64(10):3406-12. doi: 10.2337/db14-1718. Epub 2015 Jun 26. PMID 26116695
- [Result] Gastaldelli A, Gaggini M, Daniele G, Ciociaro D, Cersosimo E, Tripathy D, Triplitt C, Fox P, Musi N, DeFronzo R, Iozzo P. Exenatide improves both hepatic and adipose tissue insulin resistance: A dynamic positron emission tomography study. Hepatology. 2016 Dec;64(6):2028-2037. doi: 10.1002/hep.28827. PMID 27639082

RESULTS

PARTICIPANT FLOW:
Groups:
- OGTT-PET: Exenatide First Then Placebo: In the first study subjects received exenatide 5ug injected before OGTT-PET. In the second study (3 to 12 wk after first study), subjects received placebo injection before OGTT-PET
- OGTT-PET: Placebo First, Then Exenatide: In the first study subjects received placebo injected before OGTT-PET. In the second study (3 to 12 wk after first study), subjects received exenatide injection (5ug) before OGTT-PET
Period: Overall Study
Arm/Group | OGTT-PET: Exenatide First Then Placebo | OGTT-PET: Placebo First, Then Exenatide
Started | 11 | 4
Completed | 11 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We studied male subjects with impaired fasting glucose or newly diagnosed type 2 diabetes.
Groups:
- PET With Exenatide vs Placebo Injection: All subjects will receive the same intervention with Exenatide and placebo. Exenatide or placebo will be administered in random order, (i.e. first or second before OGTT-PET study).
  In the first study IGT male subjects will be randomized to exenatide or placebo injection before OGTT-PET study. In the second study the same subjects will receive placebo or exenatide respectively before OGTT-PET study. The results obtained after Exenatide injection will be compared with the ones obtained after injection of placebo in the same subject.
Arm/Group | PET With Exenatide vs Placebo Injection
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 29 (3)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 114 (3)
HbA1c [Mean (Standard Deviation); unit: % of total hemoglobin] | 5.6 (0.1)
2 hour plasma glucose concentration [Mean (Standard Deviation); unit: mg/dl] — glucose concentration at 2h during screening OGTT
  mg/dl | 177 (11)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Exenatide on Brain (Total Gray Matter) Glucose Metabolism
Description: To study the acute effect of exenatide on brain glucose metabolism after the glucose load. Brain glucose uptake will be determined from serial FDG PET-imaging, by using graphical methods to quantify both global and regional results. The results obtained after Exenatide injection will be compared with the ones obtained after injection of placebo in the same subject.
Time Frame: 120 minutes after exenatide or placebo injection
Population: We studied, in the same subject, the acute effect of injection of exenatide vs placebo on brain glucose metabolism (CMRglu) after the glucose load. We used FDG PET-imaging to quantify global and regional results.
Measure: Mean (Standard Error); unit: μmol/(ml*min)
Groups:
- Effect of Exenatide or Placebo on CMRglu: Brain glucose metabolism (CMRglu) during OGTT measured by PET w/ or w/out Exenatide injection
Arm/Group | Effect of Exenatide or Placebo on CMRglu
Number analyzed (Participants) | 15
μmol/(ml*min)
  total gray matter CMRglu after Exenatide | 0.14 (0.02)
  total gray matter CMRglu after Placebo | 0.10 (0.01)

2. Secondary Outcome: Effect of Exenatide on the Liver and Adipose Tissue Glucose Uptake
Description: we evaluated the acute effects of exenatide on hepatic (Hep-IR) and adipose (Adipo-IR) insulin resistance and glucose uptake.
Time Frame: 60 minutes after exenatide or placebo injection
Population: Outcome data was not collected
Arm/Group | Exenatide First, Then Placebo | Placebo First, Then Exenatide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- PET With Exenatide or Placebo Injection: This is a crossover study where all subjects received the same intervention with Exenatide and placebo, acutely in random order, (i.e. first or second before OGTT-PET study).
Arm/Group | PET With Exenatide or Placebo Injection
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Our study has several potential limitations. It included only men. During OGTT it is difficult to evaluate the separate contributions of glucose and insulin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No